CLINICAL TRIAL: NCT07301749
Title: A Prospective Multicenter Clinical Investigation Evaluating the Safety and Efficacy of the VCFix Spinal System in Stand-alone Configuration for Vertebral Augmentation (EXPAND)
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of the VCFix Spinal System for Treatment of Vertebral Compression Fractures.
Acronym: EXPAND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amber Implants B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-VS02-EU
Record Dates: First submitted 2025-05-19; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Vertebral Compression Fracture
Keywords: VCF; EXPAND; vertebral stabilization; fracture; trauma; osteoporosis; expandable implant
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VCFix Spinal System (Experimental)
  Interventions: Device: VCFix Spinal System in stand-alone configuration

INTERVENTIONS:
Device: VCFix Spinal System in stand-alone configuration — The distinguishing features of this inetrvention reside in:
  1. In situ adjustment and maintenance of the height and angle of the device that allows expansion of the fractured VB in the cranio-caudal direction to realign the vertebral endplates and correct kyphosis.
  2. The complex titanium perforated structure with optimized surface roughness that allows possible bone attachment, thereby permitting natural healing of the bone and potentially providing more stability to the device and the treated vertebra over time.
  3. The ability to likely secure and reinforce the vertebra without using PMMA bone cement, avoiding all the symptomatic and asymptomatic side effects of bone cement.
  4. The ability to connect the posterior to the anterior column of the spine through the pedicle screw component of the VCFix implant, therefore improving the biomechanical load distribution and consequently the ability to stabilize more severe fractures.

SUMMARY:
The primary objective of the EXPAND clinical investigation is to evaluate the safety and efficacy of the VCFix Spinal System for the treatment of Vertebral Compression Fractures. The study aims to demonstrate a reduction in vertebral fracture-related pain and an improvement in physical function and mobility, while ensuring the absence of (serious) adverse events ((S)AE) related to the device or procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 21 to ≤ 85 years old.
2. Single vertebral fracture which meets all of the following criteria:

   * Type A fractures from AO spine classification (compression injuries);
   * Vertebral fracture located in the thoracic and lumbar regions of the spine
   * Fracture age < 6 weeks or fractures with anatomic signs of reducibility (based on radiographic evidence as well as patient history)
   * Vertebral fracture shows an estimated height loss in the anterior or mid third of the vertebral body (VB) of at least 10% but not more than 60% based on radiographic evidence
   * Target VB has appropriate anatomy, i.e. suitable pedicle diameter, pedicle length and chord length that would allow for selection of correct implant size, as described in the IFU and based on axial MRI/CT scan before surgery
3. Subject has a NPRS back pain score of ≥5
4. Subject is a candidate for surgical intervention based on investigator opinion
5. Subject has a body Mass Index (BMI) < 35
6. Subject is mentally capable of complying with trial protocol requirements for the duration of the study
7. Subject can understand the risks and benefits of participating in the study and is able to provide written informed consent

Exclusion Criteria:

1. Neoplasms with posterior involvement and/or presence of a mass within the spinal canal
2. Non-mobile fractures (i.e., fracture is not recent (>6 weeks), bone marrow edema or fluid or empty cleft are not visible in radiographic imaging, or fracture mode does not allow for fracture reduction in craniocaudal direction).
3. Spondylolisthesis > Grade 1 at target vertebral body(s)
4. Local kyphotic angle > 30°
5. Pre-existing vertebral fracture prior to the index fracture
6. Subjects that require anterior stabilization of the index fracture
7. Fracture to the pedicle based on radiographic evaluation
8. Spinal cord compression or canal compromise requiring decompression
9. Severe back pain due to causes other than acute fracture with NPRS score>5
10. The subject has pain based on clinical diagnosis of herniated nucleus pulposus or severe spinal stenosis (progressive weakness or paralysis)
11. Pain due to any other condition that requires daily narcotic (opiates or opioids) medication
12. Pre-existing neurological deficit, radiculopathy or myelopathy
13. Pre-existing condition or significant co-morbidity:

    * Uncontrolled diabetes (HbA1c >8%)
    * Severe cardiopulmonary deficiencies
    * Any other condition that would impact study outcome in the opinion of the investigator
14. Contraindications to both MRI and radionuclide bone scan
15. Concurrent participation in another clinical study which could potentially interfere with the outcome of this study.
16. A life expectancy less than the study duration or undergoing palliative care
17. Subject non-ambulatory prior to fracture
18. Allergy to any components of the device/instruments used during the procedure
19. Active or incompletely treated infection of the vertebral column or active systemic infection, including unresolved urinary tract infection
20. Any underlying systemic bone disease other than osteoporosis (e.g., osteomalacia, osteogenesis imperfecta, Paget's disease, etc.)
21. Any evidence of alcohol or drug abuse.
22. Ongoing long-term steroid therapy (steroid dose ≥30 mg /day for >3 months)
23. The subject is currently on anti-cancer therapy or anti-HIV therapy
24. Pregnancy or subjects with child-bearing potential that are unwilling to use contraception throughout the study duration

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of more than 2 points in vertebral fracture-related pain intensity at 6 months after the index procedure compared to baseline as measured by a 11-point Numerical Pain Rating Scale (NPRS) | 6 months
Maintenance or improvement of function as measured by the 100-point Oswestry Disability Index (ODI) at 6 months compared to baseline | 6 months
Absence of serious adverse device effects (SADEs): No SADEs with causality rated as definite, monitored through 1 month post-procedure (safety) | 1 month

SECONDARY OUTCOMES:
Vertebral height restoration (anterior, midline, and posterior aspects) at PO (Post-Operative), 1Months FU, 6 Months FU and 12Months FU. | Post-Operative, 1Month FU, 6 Months FU, 12 Months FU
Kyphotic angle and Cobb angle improvement at Post-Operative, 1 Month FU, 6 Months FU and 12 Months FU. | Post-Operative, ost-Operative, 1 Month FU, 6 Months FU and 12 Months FU.
  Kyphotic angle and Cobb angle improvement
Reduction in vertebral fracture-related pain (measured by the 11-point Numerical Pain Rating Scale (NPRS)) | Discharge, 1, 3, 6 and 12 Months FU compared to baseline.
  Reduction in vertebral fracture-related pain
Improvement in function (measured by the 100-point Oswestry Disability Index (ODI)) at discharge, 1, 3, 6 and 12 months FU compared to baseline. | Discharge, 1, 3, 6 and 12 months FU
Improvement of Health-related quality of life (HRQoL) measured by EuroQol 5-Dimension Scale (EQ-5D-5L) at 1 Month, 3 Months, 6 Months and 12 Months post-procedure compared to baseline | 1 Month, 3 Months, 6 Months and 12 Months post-procedure compared to baseline
  Improvement of Health-related quality of life (HRQoL)
Device-related serious adverse events assessed at 12- and 24- months post-procedure. | 12 months FU, 24 months FU
  Device-related serious adverse events
All (per protocol reportable) adverse events assessed at 12- and 24- months post-procedure. | 12 Months FU, 24 Months FU

CONTACTS AND LOCATIONS:
Locations (3):
- Centre Hospitalier Métropole de Savoie, Chambéry, France
- Germany (2):
  - Wilhelmsburger Krankenhaus Groß-Sand, Hamburg
  - Krankenhaus Mechernich, Mechernich

IPD SHARING:
Plan to Share IPD: No